CLINICAL TRIAL: NCT04198740
Title: Proteomic and Metabolomic Lacrimal Fingerprint in Diverse Pathologies of the Ocular Surface
Acronym: EML-MSO
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université du Québec a Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: CE19.212
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye Syndrome; Infectious Keratoconjunctivitis; Mucous Membrane Pemphigoid; Allergic Conjunctivitis
Keywords: Lacrimal fingerprint; Metabolomics; Proteomics; Ocular surface
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis, Infectious; Pemphigoid, Benign Mucous Membrane; Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control group: Healthy, normal ocular surface
  Interventions: Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry
- Dry eye syndrome: Patients suffering from either:
  * Lacrimal insufficiency
  * Anterior blepharitis
  * Posterior blepharitis
  * Sjögren syndrome
  Interventions: Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry
- Allergic conjunctivitis: Patients suffering from allergic conjunctivitis
  Interventions: Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry
- Mucous membrane pemphigoid: Patients suffering from mucous membrane pemphigoid
  Interventions: Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry
- Infectious keratoconjunctivitis: Patients suffering from keratitis and/or conjunctivitis of various etiology:
  * Viral
  * Bacterial
  * Fungal
  * Acanthamoeba
  Interventions: Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry

INTERVENTIONS:
Diagnostic Test: Tear sample collection via Schirmer strip and subsequent analysis by mass spectrometry — During regular consultations at the ophthalmology department of the CHUM, eligible patients will undergo a standard 5 minute Schirmer tear test. The Schirmer strips will serve as tear samples and will be sent to UQAM's Department of chemistry for mass spectrometry analysis.

SUMMARY:
This study aims to obtain the lacrimal fingerprint for frequent pathologies of the ocular surface and establish a normative base for each of them.

DETAILED DESCRIPTION:
This is an exploratory study. The investigators aim to:

* Test and perfect a tear sample analysis technique by mass spectrometry with samples collected by Schirmer strips;
* Obtain the lacrimal fingerprint for various pathologies of the ocular surface, notably different forms of dry eye syndrome, infectious keratitis/conjunctivitis, mucous membrane pemphigoid and allergic conjunctivitis, and establish a normative base for each of them.

During regular clinics at the cornea service of the ophthalmology department of the CHUM (Centre Hospitalier de l'Université de Montréal), the investigators aim to recruit a few hundred patients with various pathologies of the ocular surface, notably different forms of dry eye syndrome, infectious keratitis/conjunctivitis, mucous membrane pemphigoid and allergic conjunctivitis, and collect a sample of their tears via Schirmer strip. A case report form will be completed for each patient, noting known ocular diagnoses and active topical ophthalmic medication. Schirmer strips will be sent in sterile tubes to UQAM (Université du Québec à Montréal)'s department of chemistry for analysis by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy corneas or suffering from one of these pathologies:

Dry eye syndrome; Infectious keratitis and/or conjunctivitis; Mucous membrane pemphigoid; Allergic conjunctivitis.

Exclusion Criteria:

* Patients younger than 18 years old;
* Patients incapable of giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients consulting at the cornea service of the ophthalmology department of the CHUM.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
To obtain the metabolomic and proteomic fingerprint of the studied ocular surface pathologies | 5 years
  Raw data will be analysed with MarkerView software by Sciex to identify specific over- or under-expressed markers in these ocular pathologies.

SECONDARY OUTCOMES:
To objectify changes in metabolomic and proteomic profile associated with topical treatments taken by participants in this study | 5 years
  Raw data will be analysed with the same software to identify specific changes in proteomic and/or metabolomic expression associated with the topical treatments taken by participants in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Robert, MD, M.Sc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - Université du Québec à Montréal (UQAM) - Department of Chemistry, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data.

REFERENCES:
- [Background] Karring H, Thogersen IB, Klintworth GK, Moller-Pedersen T, Enghild JJ. A dataset of human cornea proteins identified by Peptide mass fingerprinting and tandem mass spectrometry. Mol Cell Proteomics. 2005 Sep;4(9):1406-8. doi: 10.1074/mcp.D500003-MCP200. Epub 2005 May 23. PMID 15911533
- [Background] Elsobky S, Crane AM, Margolis M, Carreon TA, Bhattacharya SK. Review of application of mass spectrometry for analyses of anterior eye proteome. World J Biol Chem. 2014 May 26;5(2):106-14. doi: 10.4331/wjbc.v5.i2.106. PMID 24921002
- [Background] Zhou L, Zhao SZ, Koh SK, Chen L, Vaz C, Tanavde V, Li XR, Beuerman RW. In-depth analysis of the human tear proteome. J Proteomics. 2012 Jul 16;75(13):3877-85. doi: 10.1016/j.jprot.2012.04.053. Epub 2012 May 23. PMID 22634083
- [Background] Karnati R, Laurie DE, Laurie GW. Lacritin and the tear proteome as natural replacement therapy for dry eye. Exp Eye Res. 2013 Dec;117:39-52. doi: 10.1016/j.exer.2013.05.020. Epub 2013 Jun 12. PMID 23769845
- [Background] de Souza GA, Godoy LM, Mann M. Identification of 491 proteins in the tear fluid proteome reveals a large number of proteases and protease inhibitors. Genome Biol. 2006;7(8):R72. doi: 10.1186/gb-2006-7-8-R72. Epub 2006 Aug 10. PMID 16901338
- [Background] Hagan S, Martin E, Enriquez-de-Salamanca A. Tear fluid biomarkers in ocular and systemic disease: potential use for predictive, preventive and personalised medicine. EPMA J. 2016 Jul 13;7(1):15. doi: 10.1186/s13167-016-0065-3. eCollection 2016. PMID 27413414
- [Background] Willcox MDP, Argueso P, Georgiev GA, Holopainen JM, Laurie GW, Millar TJ, Papas EB, Rolland JP, Schmidt TA, Stahl U, Suarez T, Subbaraman LN, Ucakhan OO, Jones L. TFOS DEWS II Tear Film Report. Ocul Surf. 2017 Jul;15(3):366-403. doi: 10.1016/j.jtos.2017.03.006. Epub 2017 Jul 20. PMID 28736338
- [Background] Aluru SV, Agarwal S, Srinivasan B, Iyer GK, Rajappa SM, Tatu U, Padmanabhan P, Subramanian N, Narayanasamy A. Lacrimal proline rich 4 (LPRR4) protein in the tear fluid is a potential biomarker of dry eye syndrome. PLoS One. 2012;7(12):e51979. doi: 10.1371/journal.pone.0051979. Epub 2012 Dec 18. PMID 23272196
- [Background] Enriquez-de-Salamanca A, Castellanos E, Stern ME, Fernandez I, Carreno E, Garcia-Vazquez C, Herreras JM, Calonge M. Tear cytokine and chemokine analysis and clinical correlations in evaporative-type dry eye disease. Mol Vis. 2010 May 19;16:862-73. PMID 20508732
- [Background] Green-Church KB, Nichols KK, Kleinholz NM, Zhang L, Nichols JJ. Investigation of the human tear film proteome using multiple proteomic approaches. Mol Vis. 2008 Mar 7;14:456-70. PMID 18334958